CLINICAL TRIAL: NCT02618577
Title: Non-vitamin K Antagonist Oral Anticoagulants in Patients With Atrial High Rate Episodes - An Investigator-driven, Prospective, Randomised, Double-blind, Multi-centre Trial Initiated by the European Society of Cardiology and AFNET
Brief Title: Non-vitamin K Antagonist Oral Anticoagulants in Patients With Atrial High Rate Episodes
Acronym: NOAH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: following a recommendation from the data safety and monitoring board due to safety concerns and a tendency towards futility.
Sponsor: Atrial Fibrillation Network (Other)
Collaborators: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry); Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NOAH - AFNET 6; 2015-003997-33 (EudraCT Number)
Record Dates: First submitted 2015-11-27; First posted 2015-12-01 (Estimated); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Atrial High Rate Episodes
Keywords: Anticoagulation; Atrial High Rate Episodes; Atrial Fibrillation; VKA; NOAC
MeSH Terms: conditions — Atrial Fibrillation | interventions — edoxaban

STUDY DESIGN:
Intervention Model Description: Phase 3b
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Edoxaban (Experimental): Edoxaban will be applied in NOAH at the therapeutic dose approved for stroke prevention in non-valvular AF, i.e. 60 mg OD with a reduction of dose to 30 mg OD in patients with one of the following characteristics:
  Impaired renal function (CrCl 15-50 ml/min), or low body weight (≤60 kg), or patients receiving the glycoprotein-P inhibitors cyclosporin, dronedarone, erythromycin, or ketoconazole.
  Interventions: Drug: Edoxaban
- ASA or Placebo (Active Comparator): Either one tablet of ASA 100 mg plus one placebo tablet matching in colour, form and size to edoxaban 60 mg or one placebo tablet matching in colour, weight, form and size to ASA 100 mg plus one placebo tablet matching in colour, form and size to edoxaban 60 mg will be administered per day depending on the indication for use of antiplatelet therapy as assessed by the responsible investigator
  Interventions: Drug: ASA

INTERVENTIONS:
Drug: Edoxaban — Edoxaban will be applied at the therapeutic dose approved for stroke prevention in non-valvular AF
  Other Names: Lixiana; Savaysa
  Arms: Edoxaban
Drug: ASA — ASA 100 mg tablets or Placebo, based on accepted indication for the latter, including peripheral or coronary artery disease, a prior myocardial infarction, or a prior stroke.
  Other Names: ASS
  Arms: ASA or Placebo

SUMMARY:
NOAH is an investigator-initiated, prospective, parallel-group, double-blind, randomised, multi-centre trial. The objective of the trial is to demonstrate that oral anticoagulation using the NOAC edoxaban is superior to current therapy to pre-vent stroke, systemic embolism, or cardiovascular death in patients with AHRE and at least two stroke risk factors but without AF. The trial will be conducted in several European countries.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a common cause of stroke, especially ischemic stroke. So far, all available data that demonstrate a beneficial effect of oral anticoagulation for stroke prevention have been collected in populations with AF documented by conventional ECG recordings. It is well established that a large proportion of AF episodes remain undiagnosed ("silent AF"), and many of these patients present with a stroke as the first clinical sign of AF. Earlier initiation of anticoagulation could prevent such events. Continuous monitoring of atrial rhythm by implanted devices could close this diagnostic gap. Pacemakers, defibrillators, and cardiac resynchronisation devices already provide automated algorithms alerting to the occurrence of highly organised atrial tachyarrhythmia episodes, also called "subclinical atrial fibrillation" or, more commonly, "atrial high rate episodes" (AHRE). Data from large prospectively followed patient cohorts demonstrated that stroke rate is increased in patients with AHRE. A sizeable portion of these patients develops clinically detected AF over time. In these patients, AHRE can be considered as an early manifestation of paroxysmal AF. A few AHRE patients do not develop clinically overt AF, and the absolute stroke rates are lower in patients with AHRE when compared to stroke rates in patients with clinically diagnosed AF. In light of the bleeding complications associated with oral anticoagulant therapy, there is thus uncertainty about the optimal antithrombotic therapy in patients with AHREs.

The Non-vitamin K antagonist Oral anticoagulants (NOACs) provide similar or slightly better stroke prevention, and appear slightly safer compared to vitamin K antagonists (VKAs). In addition, no individual therapy adjustment of NOACs has to be performed. Edoxaban, a newly introduced NOAC, at a dose regime of 60 mg once daily (OD) has a favourable profile compared to dose-adjusted VKA therapy: In the ENGAGE-TIMI 48 trial, edoxaban prevented strokes at least as effectively as VKA therapy but caused less major bleeding events than VKA therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pacemaker, defibrillator or insertable cardiac monitor implanted for any reason with feature of detection of AHRE, implanted at least 2 months prior to randomisation
* AHRE detection feature activated for adequate detection of AHRE (refer to Appendix XIII)
* AHRE (≥ 170 bpm atrial rate and ≥ 6 min duration) documented by the implanted device via its atrial lead and stored digitally. Any AHRE episode recorded is potentially eligible, but AHRE episodes detected in the first 2 months after implantation of a new device involving placement or repositioning of atrial electrodes are not eligible. AHRE episodes recorded in the first two months after a simple "box change" operation, i.e. exchange of a pacemaker or defibrillator device without exchange or repositioning of atrial electrodes, are eligible
* Provision of signed informed consent
* Age ≥ 65 years

In addition, at least one of the following cardiovascular conditions leading to a modified CHA2DS2VASc score of 2 or more:

* Age ≥ 75 years
* Heart failure (clinically overt or LVEF < 45%)
* Arterial hypertension (chronic treatment for hypertension, estimated need for continuous antihyper-tensive therapy or resting blood pressure > 145/90 mmHg)
* Diabetes mellitus
* Prior stroke or transient ischemic attack (TIA)
* Vascular disease (previous myocardial infarction, peripheral, carotid/cerebral, or aortic plaques on transesophageal echocardiogram [TEE])
* Provision of signed informed consent

Exclusion Criteria:

* Any disease that limits life expectancy to less than 1 year
* Participation in another controlled clinical trial, either within the past two months or still ongoing
* Previous participation in the present trial NOAH - AFNET 6
* Drug abuse or clinically manifest alcohol abuse
* Any history of overt AF or atrial flutter
* Indication for oral anticoagulation (e.g. deep venous thrombosis)
* Contraindication for oral anticoagulation in general
* Contraindication for edoxaban as stated in the current SmPC
* Indication for long-term antiplatelet therapy other than acetylsalicylic acid or a need for treatment with any antiplatelet agent in addition to edoxaban, especially dual antiplatelet therapy (DAPT). Patients with a transient requirement for DAPT (e.g. after receiving a stent) will be eligible when the need for DAPT is no longer present
* Acute coronary syndrome, coronary revascularisation (PCI or bypass surgery), or overt stroke within 30 days prior to randomisation
* End stage renal disease (creatinine clearance (CrCl) < 15 ml/min as calculated by the Cockcroft-Gault method)
* All persons exempt from participation in a clinical trial by law

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2608 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paulus Kirchhof, Prof. Dr., Principal Investigator — University Clinic of Hamburg-Eppendorf, Hamburg, Germany
Locations (18):
- Several Sites, Multiple Locations, Austria
- Several Sites, Multiple Locations, Belgium
- Several, Multiple Locations, Bulgaria
- Several, Multiple Locations, Czechia
- Several, Multiple Locations, Denmark
- Several, Multiple Locations, France
- Several Sites, Multiple Locations, Germany
- Several, Multiple Locations, Greece
- Several, Multiple Locations, Hungary
- Several, Multiple Locations, Italy
- Several, Multiple Locations, Netherlands
- Several, Multiple Locations, Poland
- Several, Multiple Locations, Portugal
- Several, Multiple Locations, Romania
- Several, Multiple Locations, Spain
- Several, Multiple Locations, Sweden
- Several, Multiple Locations, Ukraine
- Several, Multiple Locations, United Kingdom

REFERENCES:
- [Background] Bertaglia E, Blank B, Blomstrom-Lundqvist C, Brandes A, Cabanelas N, Dan GA, Dichtl W, Goette A, de Groot JR, Lubinski A, Marijon E, Merkely B, Mont L, Piorkowski C, Sarkozy A, Sulke N, Vardas P, Velchev V, Wichterle D, Kirchhof P. Atrial high-rate episodes: prevalence, stroke risk, implications for management, and clinical gaps in evidence. Europace. 2019 Oct 1;21(10):1459-1467. doi: 10.1093/europace/euz172. PMID 31377792
- [Background] Kirchhof P, Blank BF, Calvert M, Camm AJ, Chlouverakis G, Diener HC, Goette A, Huening A, Lip GYH, Simantirakis E, Vardas P. Probing oral anticoagulation in patients with atrial high rate episodes: Rationale and design of the Non-vitamin K antagonist Oral anticoagulants in patients with Atrial High rate episodes (NOAH-AFNET 6) trial. Am Heart J. 2017 Aug;190:12-18. doi: 10.1016/j.ahj.2017.04.015. Epub 2017 May 3. PMID 28760205
- [Derived] Kirchhof P, Toennis T, Goette A, Camm AJ, Diener HC, Becher N, Bertaglia E, Blomstrom Lundqvist C, Borlich M, Brandes A, Cabanelas N, Calvert M, Chlouverakis G, Dan GA, de Groot JR, Dichtl W, Kravchuk B, Lubinski A, Marijon E, Merkely B, Mont L, Ozga AK, Rajappan K, Sarkozy A, Scherr D, Sznajder R, Velchev V, Wichterle D, Sehner S, Simantirakis E, Lip GYH, Vardas P, Schotten U, Zapf A; NOAH-AFNET 6 Investigators; NOAH-AFNET6 sites and investigators. Anticoagulation with Edoxaban in Patients with Atrial High-Rate Episodes. N Engl J Med. 2023 Sep 28;389(13):1167-1179. doi: 10.1056/NEJMoa2303062. Epub 2023 Aug 25. PMID 37622677
- See also: NOAH Trial — https://www.kompetenznetz-vorhofflimmern.de/de/forschung/laufende-studien-und-projekte/noah-afnet-6

RESULTS

PARTICIPANT FLOW:
Groups:
- Edoxaban: Edoxaban will be applied in NOAH at the therapeutic dose approved for stroke prevention in non-valvular AF, i.e. 60 mg OD with a reduction of dose to 30 mg OD in patients with one of the following characteristics:
  Impaired renal function (CrCl 15-50 ml/min), or low body weight (≤60 kg), or patients receiving the glycoprotein-P inhibitors cyclosporin, dronedarone, erythromycin, or ketoconazole.
  Edoxaban: Edoxaban will be applied at the therapeutic dose approved for stroke prevention in non-valvular AF, i.e. 60 mg OD with a reduction of dose to 30 mg OD in patients with one of the following characteristics:
  Impaired renal function (CrCl 15-50 ml/min), or low body weight (≤60 kg), or patients receiving the glycoprotein-P inhibitors cyclosporin, dronedarone, erythromycin, or ketoconazole.
- ASA or Placebo: Either one tablet of ASA 100 mg plus one placebo tablet matching in colour, form and size to edoxaban 60 mg or one placebo tablet matching in colour, weight, form and size to ASA 100 mg plus one placebo tablet matching in colour, form and size to edoxaban 60 mg will be administered per day depending on the indication for use of antiplatelet therapy as assessed by the responsible investigator
  ASA: ASA 100 mg tablets or Placebo, based on accepted indication for the latter, including peripherial or coronary artery disease, a prior myocardial infarction, or a prior stroke.
Period: Overall Study
Arm/Group | Edoxaban | ASA or Placebo
Started | 1306 | 1302
Completed | 500 | 472
Not Completed | 806 | 830

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Edoxaban | ASA or Placebo | Total
Number analyzed (Participants) | 1270 | 1264 | 2534
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.4 (6.5) | 77.5 (6.8) | 77.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 469 | 478 | 947
  Male | 801 | 786 | 1587
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Romania | 7 | 7 | 14
  Hungary | 35 | 35 | 70
  Czechia | 6 | 6 | 12
  Ukraine | 179 | 172 | 351
  United Kingdom | 76 | 80 | 156
  Portugal | 13 | 12 | 25
  Spain | 176 | 177 | 353
  Greece | 4 | 3 | 7
  Austria | 108 | 113 | 221
  Netherlands | 22 | 28 | 50
  Sweden | 9 | 7 | 16
  Belgium | 15 | 8 | 23
  Poland | 137 | 135 | 272
  Denmark | 11 | 7 | 18
  Italy | 82 | 76 | 158
  Bulgaria | 9 | 12 | 21
  France | 41 | 41 | 82
  Germany | 340 | 345 | 685

OUTCOME MEASURES:

1. Primary Outcome: Composite of Stroke, Systemic Embolism, or Cardiovascular Death
Description: Time from randomisation to the first occurrence of stroke, systemic embolism, or cardiovascular death; incidence of first occurence of outcome measure.
Time Frame: 28 months
Population: The primary analysis is in the modified intention-to-treat population, consisting of all randomised patients with a qualifying AHRE and intake of at least one dose of study drug.
Measure: Number; unit: number of new events per 100 pat.-years
Units Other Than Participants: patient-years
Arm/Group | Edoxaban | ASA or Placebo
Number analyzed (Participants) | 1270 | 1264
Number analyzed (patient-years) | 2556 | 2494
number of new events per 100 pat.-years | 3.3 | 4.0
Statistical Analysis 1: Comparison: Edoxaban vs ASA or Placebo; Test type: Superiority; p = 0.15, Cause-spec. Cox Proport. Hazard model; adjusted cause-specific hazard ratio = 0.81, 95% CI 2-sided [0.6 to 1.08]

2. Secondary Outcome: Components of the Primary Outcome, Stroke
Description: Time from randomisation to the first occurrence of ischemic stroke; incidence of first occurence of outcome measure.
Time Frame: 28 months
Measure: Number; unit: number of new events per 100 pat.-years
Units Other Than Participants: patient-years
Arm/Group | Edoxaban | ASA or Placebo
Number analyzed (Participants) | 1270 | 1264
Number analyzed (patient-years) | 2572 | 2518
number of new events per 100 pat.-years | 0.9 | 1.1
Statistical Analysis 1: Comparison: Edoxaban vs ASA or Placebo; Test type: Superiority; adjusted cause-specific hazard ratio = 0.79, 95% CI 2-sided [0.45 to 1.39]

3. Secondary Outcome: Major Adverse Cardiac Events (MACEs: Cardiac Death, Myocardial Infarction, Acute Coronary Syndrome (ACS)
Description: PCI, CABG
Time Frame: 28 months
Measure: Number; unit: number of new events per 100 pat.-years
Units Other Than Participants: patient-years
Arm/Group | Edoxaban | ASA or Placebo
Number analyzed (Participants) | 1270 | 1264
Number analyzed (patient-years) | 2532 | 2484
number of new events per 100 pat.-years | 3.6 | 4.1
Statistical Analysis 1: Comparison: Edoxaban vs ASA or Placebo; Test type: Superiority; adjusted cause-specific hazard ratio = 0.89, 95% CI 2-sided [0.67 to 1.18]

4. Secondary Outcome: All-cause Death
Description: All-cause death
Time Frame: 28 months
Measure: Number; unit: number of new events per 100 pat.-years
Units Other Than Participants: patient-years
Arm/Group | Edoxaban | ASA or Placebo
Number analyzed (Participants) | 1270 | 1264
Number analyzed (patient-years) | 2595 | 2539
number of new events per 100 pat.-years | 4.3 | 3.7
Statistical Analysis 1: Comparison: Edoxaban vs ASA or Placebo; Test type: Superiority; p = 0.28, Cause-spec. Cox Proport. Hazard model; adjusted cause-specific hazard ratio = 1.16, 95% CI 2-sided [0.88 to 1.53]

5. Secondary Outcome: Major Bleeding Events
Description: according to the International Society on Thrombosis and Haemostasis (ISTH) definitions
Time Frame: 28 months
Measure: Number; unit: number of new events per 100 pat.-years
Units Other Than Participants: patient-years
Arm/Group | Edoxaban | ASA or Placebo
Number analyzed (Participants) | 1270 | 1264
Number analyzed (patient-years) | 2533 | 2507
number of new events per 100 pat.-years | 2.1 | 1.0
Statistical Analysis 1: Comparison: Edoxaban vs ASA or Placebo; Test type: Superiority; p = 0.002, Cause-spec. Cox Proport. Hazard model; adjusted cause-specific hazard ratio = 2.1, 95% CI 2-sided [1.3 to 3.38]

6. Secondary Outcome: Quality of Life Changes at 12 and 24 Months Compared to Baseline
Description: Adjusted mean change from baseline at 12 and 24 months of Quality of life as assessed by the EuroQol Group 5-Dimension 5-Level questionnaire (EQ-5D-5L): The resulting score of the UK index ranges from 1 (for the best state) to - 0.285 (for the worst state), with 5.1% of the states valued as worse than dead. EQ5D- VAS: visual-analogue scale (0 worst to 100 best).
  Subscales of the UK index score were combined by adding up EQ-5D-5L index values with STATA using the English (ENG) Devlin value set, Version 1.1 (Updated 01/12/2020).
  Karnofsky Performance Scale is an 11-point scale from 0 to 100 (0 worst to 100 best).
Time Frame: Baseline, 12 months and 24 months.
Measure: Number (95% Confidence Interval); unit: adjusted mean change from baseline
Arm/Group | Edoxaban | ASA or Placebo
Number analyzed (Participants) | 1270 | 1264
adjusted mean change from baseline
  EQ-5D-5L UK Index to FU12 | -0.01 [-0.03 to 0] | -0.01 [-0.02 to 0.01]
  EQ-5D-5L UK Index to FU24 | -0.04 [-0.05 to -0.02] | -0.03 [-0.05 to -0.02]
  EQ-5D-5L VAS to FU12 | -0.75 [-2.08 to 0.57] | -0.71 [-2.06 to 0.64]
  EQ-5D-5L VAS to FU24 | -1.72 [-3.18 to -0.27] | -1.68 [-3.16 to 0.20]
  Karnofsky score to FU12 | -1.14 [-1.98 to -0.31] | -1.41 [-2.26 to -0.57]
  Karnofsky score to FU24 | -2.28 [-3.23 to -1.33] | -2.55 [-3.50 to -1.59]
Statistical Analysis 1: Comparison: Edoxaban vs ASA or Placebo; EQ-5D-5L UK Index; Test type: Superiority; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.02 to 0.01] — Estimation Parameter: baseline adjusted trial-group specific effect estimates (mean difference)
Statistical Analysis 2: Comparison: Edoxaban vs ASA or Placebo; EQ-5D-5L VAS, FU 24months; Test type: Superiority; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-1.46 to 1.38] — Estimation Parameter: baseline adjusted trial-group specific effect estimates (mean difference)
Statistical Analysis 3: Comparison: Edoxaban vs ASA or Placebo; Karnofsky score; Test type: Superiority; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.56 to 1.09] — Estimation Parameter: baseline adjusted trial-group specific effect estimates (mean difference)

7. Secondary Outcome: Patient Satisfaction at 12 and 24 Months Compared to Baseline
Description: Adjusted change from baseline at 12 and 24 months measured by the Perception of Anticoagulant Treatment Questionnaire: For convenience score, a 0 - 100 scale; for satisfaction score a 0 - 100 scale; for both scores, the higher the score, the higher the convenience/satisfaction.
Time Frame: Baseline, 12 months and 24 months.
Measure: Number (95% Confidence Interval); unit: scores on a scale (with 95% Confidence I
Arm/Group | Edoxaban | ASA or Placebo
Number analyzed (Participants) | 1270 | 1264
scores on a scale (with 95% Confidence I
  PACT-Q convenience to FU12 | 0.84 [-0.26 to 1.93] | 0.96 [-0.14 to 2.05]
  PACT-Q convenience to FU24 | 1.35 [0.2 to 2.49] | 1.47 [0.32 to 2.61]
  PACT-Q satisfaction to FU12 | 2.97 [1.36 to 4.57] | 4.01 [2.39 to 5.62]
  PACT-Q satisfaction to FU24 | 3.80 [2.12 to 5.48] | 4.84 [3.15 to 6.52]
Statistical Analysis 1: Comparison: Edoxaban vs ASA or Placebo; PACT-Q convenience; Test type: Superiority; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-1.12 to 0.87] — Estimation Parameter: baseline adjusted trial-group specific effect estimates (mean difference)
Statistical Analysis 2: Comparison: Edoxaban vs ASA or Placebo; PACT-Q satisfaction; Test type: Superiority; Mean Difference (Final Values) = -1.04, 95% CI 2-sided [-2.60 to 0.52] — Estimation Parameter: baseline adjusted trial-group specific effect estimates (mean difference)

8. Secondary Outcome: Cost Effectiveness and Health Resource Utilisation
Description: estimated by quantification of relevant events, interventions, nights spent in hospital and cardiovascular therapies
Time Frame: 28 months
Reporting Status: Not Posted

9. Secondary Outcome: Autonomy Status
Description: Autonomy status only in patients with stroke during study participation, assessed at 24 month by modified Rankin scale. (Score ranges from 1 to 8, a higher score indicates a higher grade of disability)
Time Frame: Baseline and 24 months
Population: MoCA Stroke Severity in patients with a stroke estimated by the Modified Rankin Scale at FU24.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Edoxaban | ASA or Placebo
Number analyzed (Participants) | 10 | 14
Scores on a scale | 3.0 [2.0 to 3.0] | 2.5 [2.0 to 3.0]

10. Secondary Outcome: Components of the Primary Outcome, Systemic Embolism
Description: Time from randomisation to the first occurrence of systemic embolism; incidence of first occurence of outcome measure.
Time Frame: 28 months
Measure: Number; unit: number of new events per 100 pat.-years
Units Other Than Participants: patient-years
Arm/Group | Edoxaban | ASA or Placebo
Number analyzed (Participants) | 1270 | 1264
Number analyzed (patient-years) | 2578 | 2514
number of new events per 100 pat.-years | 0.5 | 1.1
Statistical Analysis 1: Comparison: Edoxaban vs ASA or Placebo; Test type: Superiority; adjusted cause-specific hazard ratio = 0.51, 95% CI 2-sided [0.27 to 0.96]

11. Secondary Outcome: Components of the Primary Outcome, Cardiovascular Death
Description: Time from randomisation to the first occurrence of cardiovascular death; incidence of first occurence of outcome measure.
Time Frame: 28 months
Measure: Number; unit: number of new events per 100 pat.-years
Units Other Than Participants: patient-years
Arm/Group | Edoxaban | ASA or Placebo
Number analyzed (Participants) | 1270 | 1264
Number analyzed (patient-years) | 2595 | 2539
number of new events per 100 pat.-years | 2.0 | 2.2
Statistical Analysis 1: Comparison: Edoxaban vs ASA or Placebo; Test type: Superiority; adjusted cause-specific hazard ratio = 0.90, 95% CI 2-sided [0.62 to 1.31]

ADVERSE EVENTS:
Time Frame: (S)AEs were collected during a median follow-up time of 21 months after the baseline visit for all patients until the trial was terminated, i.e. (S)AEs were collected through study completion. (S)AEs were collected on a 6 monthly basis after baseline visit. After the announcement of early termination of the trial due to safety reasons and futility, a final visit was conducted within 3 months for all active patients including a final (Serious) Adverse Event assessment.
Description: Following the patient's randomisation in the study, all AEs, whether related or not related to study drug, had to be collected. However, within the context of the NOAH - AFNET 6 trial, no specific AEs and/or laboratory abnormalities are being considered as critical to safety evaluations. Thus, reporting of AEs not fulfilling any criteria of seriousness is not time critical. All-cause mortality was only assessed for mITT population, other AEs in ITT population.
Arm/Group | Edoxaban | ASA or Placebo
All-Cause Mortality (participants affected / at risk) | 142/1306 | 125/1302
Serious Adverse Events (participants affected / at risk) | 498/1306 | 467/1302
Other Adverse Events (participants affected / at risk) | 718/1306 | 662/1302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edoxaban (N=1306) | ASA or Placebo (N=1302)
Anaemia (Blood and lymphatic system disorders) | 44 (55) | 16 (26)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Paratracheal lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 3 (3) | 9 (9)
Acute myocardial infarction (Cardiac disorders) | 14 (20) | 19 (21)
Angina pectoris (Cardiac disorders) | 14 (17) | 11 (11)
Angina unstable (Cardiac disorders) | 2 (2) | 3 (3)
Aortic valve stenosis (Cardiac disorders) | 4 (5) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 38 (50) | 39 (51)
Atrial flutter (Cardiac disorders) | 6 (7) | 11 (11)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac amyloidosis (Cardiac disorders) | 0 (0) | 1 (3)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 93 (145) | 90 (131)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 6 (6) | 6 (6)
Coronary artery disease (Cardiac disorders) | 7 (7) | 8 (8)
Dilated cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 3 (4) | 3 (4)
Mitral valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 5 (5) | 6 (6)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 4 (4) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 2 (3)
Ventricular tachycardia (Cardiac disorders) | 5 (5) | 4 (5)
Haemophilia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 4 (5) | 4 (5)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Amaurosis fugax (Eye disorders) | 4 (4) | 0 (0)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 3 (3)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Retinal vein thrombosis (Eye disorders) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Visual field defect (Eye disorders) | 0 (0) | 1 (1)
Vitreoretinal traction syndrome (Eye disorders) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 5 (5)
Diverticulum (Gastrointestinal disorders) | 4 (4) | 6 (6)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 4 (4) | 3 (3)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastritis (Gastrointestinal disorders) | 5 (5) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastritis haemorrhagic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 50 (66) | 19 (23)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 6 (6) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 2 (2)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 3 (3) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 3 (4)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 1 (1)
Melaena (Gastrointestinal disorders) | 4 (4) | 4 (4)
Mesenteric artery embolism (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal mucosa erythema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 4 (6) | 3 (3)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Proctitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 4 (4) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 2 (2) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Volvulus of small bowel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 4 (4) | 3 (3)
Cardiac death (General disorders) | 21 (21) | 22 (22)
Chest pain (General disorders) | 5 (5) | 4 (4)
Death (General disorders) | 103 (103) | 87 (88)
Gait disturbance (General disorders) | 3 (3) | 0 (0)
General physical health deterioration (General disorders) | 2 (3) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Multimorbidity (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 2 (2)
Non-cardiac chest pain (General disorders) | 6 (6) | 5 (5)
Oedema (General disorders) | 0 (0) | 1 (2)
Oedema peripheral (General disorders) | 2 (2) | 2 (2)
Pacemaker generated arrhythmia (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Puncture site haemorrhage (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 4 (4)
Sudden cardiac death (General disorders) | 18 (18) | 15 (15)
Systemic inflammatory response syndrome (General disorders) | 2 (2) | 0 (0)
Ulcer (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 6 (7) | 3 (3)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary tract disorder (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 3 (3) | 3 (3)
Cholecystitis acute (Hepatobiliary disorders) | 8 (8) | 5 (5)
Cholelithiasis (Hepatobiliary disorders) | 5 (5) | 3 (3)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (2)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 2 (2) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (2)
Post cholecystectomy syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 2 (2)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 2 (2)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Brain abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 3 (3)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 2 (2)
Diverticulitis (Infections and infestations) | 6 (6) | 4 (4)
Emphysematous pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 1 (1)
Endocarditis (Infections and infestations) | 2 (2) | 3 (3)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 3 (5) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastric ulcer helicobacter (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 3 (3) | 0 (0)
Groin abscess (Infections and infestations) | 2 (2) | 1 (1)
Hepatic cyst infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis E (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 4 (4) | 7 (8)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 5 (5)
Mediastinal abscess (Infections and infestations) | 0 (0) | 1 (1)
Myelitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0)
Pancreatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Papilloma viral infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 58 (74) | 56 (61)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 6 (7) | 3 (3)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 9 (9)
Septic shock (Infections and infestations) | 9 (9) | 5 (5)
Streptococcal endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Superinfection (Infections and infestations) | 1 (1) | 0 (0)
Superinfection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 23 (25) | 19 (21)
Urosepsis (Infections and infestations) | 3 (3) | 7 (7)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Accident at home (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 16 (17) | 20 (23)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Femur fracture (Injury, poisoning and procedural complications) | 9 (9) | 10 (10)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Immunisation reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 3 (4) | 7 (7)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nasal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 3 (3) | 6 (7)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Reactive gastropathy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Scrotal haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Angiocardiogram (Investigations) | 20 (22) | 26 (26)
Angiogram (Investigations) | 1 (1) | 4 (4)
Arteriogram carotid (Investigations) | 0 (0) | 1 (1)
Aspiration joint (Investigations) | 1 (1) | 1 (1)
Aspiration pleural cavity (Investigations) | 0 (0) | 1 (1)
Biopsy (Investigations) | 4 (4) | 1 (1)
Biopsy adrenal gland (Investigations) | 1 (1) | 0 (0)
Biopsy bladder (Investigations) | 1 (1) | 1 (1)
Biopsy heart (Investigations) | 1 (1) | 0 (0)
Biopsy kidney (Investigations) | 1 (1) | 0 (0)
Biopsy lung (Investigations) | 2 (2) | 0 (0)
Biopsy lymph gland (Investigations) | 1 (1) | 1 (1)
Biopsy pericardium (Investigations) | 1 (1) | 0 (0)
Biopsy prostate (Investigations) | 1 (1) | 0 (0)
Biopsy skin (Investigations) | 0 (0) | 1 (1)
Capsule endoscopy (Investigations) | 1 (1) | 1 (1)
Cardiac electrophysiologic study (Investigations) | 1 (1) | 0 (0)
Cardiac pacemaker evaluation (Investigations) | 0 (0) | 1 (1)
Catheterisation cardiac (Investigations) | 2 (2) | 0 (0)
Colonoscopy (Investigations) | 37 (45) | 20 (21)
Coronavirus test positive (Investigations) | 34 (41) | 36 (37)
Cystoscopy (Investigations) | 4 (4) | 0 (0)
Diagnostic procedure (Investigations) | 40 (48) | 16 (18)
Electrocardiogram ambulatory (Investigations) | 1 (1) | 0 (0)
Endoscopic retrograde cholangiopancreatography (Investigations) | 14 (17) | 6 (6)
Endoscopy small intestine (Investigations) | 1 (1) | 0 (0)
Endoscopy upper gastrointestinal tract (Investigations) | 54 (64) | 23 (27)
Human rhinovirus test positive (Investigations) | 1 (1) | 0 (0)
Mediastinoscopy (Investigations) | 1 (1) | 0 (0)
Oesophageal manometry (Investigations) | 0 (0) | 1 (1)
Oesophagogastroduodenoscopy (Investigations) | 1 (1) | 0 (0)
Paranasal biopsy (Investigations) | 1 (1) | 0 (0)
Pneumovirus test positive (Investigations) | 1 (1) | 0 (0)
Sleep study (Investigations) | 1 (1) | 0 (0)
Ureteroscopy abnormal (Investigations) | 0 (0) | 1 (1)
Venogram (Investigations) | 1 (1) | 0 (0)
Viral test negative (Investigations) | 95 (130) | 93 (122)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 6 (7) | 7 (8)
Diabetes mellitus (Metabolism and nutrition disorders) | 4 (5) | 2 (3)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (3) | 3 (3)
Gout (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 3 (4)
Iron deficiency (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 (8) | 10 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 0 (0)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 2 (4)
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (14) | 2 (2)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (6) | 0 (0)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (5) | 1 (2)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (11) | 6 (9)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to the mediastinum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 2 (2)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (7) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (4)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pleural mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 3 (4)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Renal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 2 (3)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (4)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 3 (3)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 2 (2) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 2 (2)
Dementia Alzheimer's type (Nervous system disorders) | 1 (2) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1)
Embolic stroke (Nervous system disorders) | 7 (7) | 9 (9)
Epilepsy (Nervous system disorders) | 4 (4) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (3)
Ischaemic stroke (Nervous system disorders) | 25 (25) | 29 (30)
Lacunar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 2 (2)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0)
Paraplegia (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 2 (2) | 2 (2)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 2 (3) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 3 (3) | 4 (4)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 4 (4)
Syncope (Nervous system disorders) | 9 (11) | 9 (9)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 6 (7) | 5 (5)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Device inappropriate shock delivery (Product Issues) | 1 (1) | 0 (0)
Device lead issue (Product Issues) | 3 (3) | 4 (4)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Lead dislodgement (Product Issues) | 1 (1) | 4 (4)
Undersensing (Product Issues) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 0 (0)
Chronic idiopathic pain syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Disturbance in social behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Drug dependence (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Suicide attempt (Psychiatric disorders) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 14 (14) | 13 (14)
Bladder disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 6 (7)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 9 (13) | 8 (10)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 6 (6) | 5 (6)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal pelvis fistula (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urethral haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 2 (2) | 2 (2)
Urinary retention (Renal and urinary disorders) | 4 (4) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Genital lesion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 8 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cystic lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 8 (8)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 8 (10)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 10 (10)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 7 (7)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 4 (6) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Abdominal cavity drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Abdominal wall operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Abscess drainage (Surgical and medical procedures) | 1 (1) | 1 (1)
Amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Anal lesion excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Aneurysm repair (Surgical and medical procedures) | 1 (1) | 1 (1)
Angioplasty (Surgical and medical procedures) | 5 (7) | 5 (5)
Aortic aneurysm repair (Surgical and medical procedures) | 4 (4) | 0 (0)
Aortic bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic valve replacement (Surgical and medical procedures) | 3 (3) | 2 (2)
Appendicectomy (Surgical and medical procedures) | 2 (2) | 3 (3)
Arterial aneurysm repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Arterial stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Arteriovenous fistula operation (Surgical and medical procedures) | 0 (0) | 1 (2)
Arthrodesis (Surgical and medical procedures) | 0 (0) | 1 (1)
Atrial appendage closure (Surgical and medical procedures) | 4 (4) | 1 (1)
Bile duct stent insertion (Surgical and medical procedures) | 1 (1) | 1 (1)
Bile duct stent removal (Surgical and medical procedures) | 1 (1) | 1 (1)
Biliary catheter insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Bladder catheter removal (Surgical and medical procedures) | 2 (2) | 0 (0)
Bladder catheter temporary (Surgical and medical procedures) | 1 (1) | 1 (1)
Bladder catheterisation (Surgical and medical procedures) | 3 (3) | 1 (1)
Bladder neoplasm surgery (Surgical and medical procedures) | 3 (3) | 0 (0)
Bladder polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Brachytherapy (Surgical and medical procedures) | 1 (1) | 1 (2)
Breast conserving surgery (Surgical and medical procedures) | 0 (0) | 2 (2)
Breast prosthesis removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Bunion operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Bursa removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Cancer surgery (Surgical and medical procedures) | 3 (3) | 3 (3)
Cardiac ablation (Surgical and medical procedures) | 15 (16) | 15 (15)
Cardiac pacemaker adjustment (Surgical and medical procedures) | 1 (1) | 3 (3)
Cardiac pacemaker insertion (Surgical and medical procedures) | 3 (3) | 1 (1)
Cardiac pacemaker removal (Surgical and medical procedures) | 2 (2) | 4 (4)
Cardiac pacemaker replacement (Surgical and medical procedures) | 38 (39) | 57 (58)
Cardiac resynchronisation therapy (Surgical and medical procedures) | 19 (20) | 13 (14)
Cardioversion (Surgical and medical procedures) | 21 (29) | 21 (22)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Cataract operation (Surgical and medical procedures) | 0 (0) | 2 (2)
Central venous catheter removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Central venous catheterisation (Surgical and medical procedures) | 1 (1) | 1 (1)
Chemotherapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 11 (11) | 6 (6)
Cholelithotomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Circumcision (Surgical and medical procedures) | 1 (1) | 0 (0)
Colectomy (Surgical and medical procedures) | 8 (9) | 3 (3)
Colostomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Coronary angioplasty (Surgical and medical procedures) | 3 (3) | 2 (3)
Coronary arterial stent insertion (Surgical and medical procedures) | 29 (32) | 27 (30)
Coronary artery bypass (Surgical and medical procedures) | 5 (5) | 4 (4)
Corpora cavernosa surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Craniectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cyst drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Cytoreductive surgery (Surgical and medical procedures) | 0 (0) | 2 (2)
Debridement (Surgical and medical procedures) | 1 (1) | 1 (1)
Duodenal sphincterotomy (Surgical and medical procedures) | 2 (2) | 0 (0)
Duodenectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Ear tube insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Electrocoagulation (Surgical and medical procedures) | 1 (1) | 0 (0)
Endarterectomy (Surgical and medical procedures) | 3 (3) | 1 (1)
Eventration repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Eyelid operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Foot amputation (Surgical and medical procedures) | 1 (1) | 1 (1)
Gastrectomy (Surgical and medical procedures) | 2 (3) | 1 (1)
Gastrointestinal endoscopic therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastrostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Glossectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Haematoma evacuation (Surgical and medical procedures) | 0 (0) | 1 (1)
Haemodialysis (Surgical and medical procedures) | 1 (1) | 1 (1)
Haemorrhoid operation (Surgical and medical procedures) | 2 (2) | 1 (1)
Hernia repair (Surgical and medical procedures) | 1 (2) | 3 (3)
High frequency ablation (Surgical and medical procedures) | 2 (2) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 16 (17) | 11 (11)
Hip surgery (Surgical and medical procedures) | 2 (2) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 3 (3) | 2 (2)
Ileostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Immunochemotherapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Infiltration anaesthesia (Surgical and medical procedures) | 0 (0) | 1 (1)
Inguinal hernia repair (Surgical and medical procedures) | 3 (3) | 4 (4)
Internal fixation of fracture (Surgical and medical procedures) | 9 (10) | 9 (9)
Intestinal operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Intra-aortic balloon placement (Surgical and medical procedures) | 1 (1) | 0 (0)
Intraocular lens implant (Surgical and medical procedures) | 0 (0) | 1 (1)
Jejunectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Joint fluid drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 6 (6) | 6 (6)
Knee operation (Surgical and medical procedures) | 1 (1) | 4 (4)
Laparoscopic surgery (Surgical and medical procedures) | 2 (2) | 1 (1)
Laparotomy (Surgical and medical procedures) | 5 (5) | 1 (1)
Large intestinal polypectomy (Surgical and medical procedures) | 3 (3) | 2 (2)
Laryngeal operation (Surgical and medical procedures) | 1 (1) | 1 (1)
Laryngeal prosthesis placement (Surgical and medical procedures) | 0 (0) | 1 (1)
Laryngectomy (Surgical and medical procedures) | 2 (2) | 1 (1)
Lesion excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Limb amputation (Surgical and medical procedures) | 2 (2) | 1 (1)
Lithotripsy (Surgical and medical procedures) | 0 (0) | 1 (1)
Liver ablation (Surgical and medical procedures) | 1 (3) | 0 (0)
Liver operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Lung lobectomy (Surgical and medical procedures) | 3 (3) | 0 (0)
Lymphadenectomy (Surgical and medical procedures) | 1 (1) | 3 (3)
Mammoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Medical device implantation (Surgical and medical procedures) | 1 (1) | 0 (0)
Meningioma surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Mitral valve repair (Surgical and medical procedures) | 3 (4) | 3 (3)
Neck dissection (Surgical and medical procedures) | 0 (0) | 1 (1)
Nephrectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Nephrostomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Oesophageal dilation procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Oesophageal prosthesis insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Orthopaedic procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Pancreaticoduodenectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Paracentesis (Surgical and medical procedures) | 1 (1) | 0 (0)
Parathyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Parotidectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Pelvic operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Percutaneous coronary intervention (Surgical and medical procedures) | 28 (33) | 36 (39)
Pericardial drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Peripheral artery angioplasty (Surgical and medical procedures) | 4 (4) | 3 (3)
Peripheral artery bypass (Surgical and medical procedures) | 1 (2) | 1 (1)
Peripheral artery stent insertion (Surgical and medical procedures) | 3 (3) | 4 (4)
Peripheral nerve destruction (Surgical and medical procedures) | 1 (1) | 0 (0)
Pharyngeal fistula repair (Surgical and medical procedures) | 1 (2) | 0 (0)
Pharyngeal operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Pleurectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Polypectomy (Surgical and medical procedures) | 2 (2) | 1 (1)
Positive airway pressure therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Proctectomy (Surgical and medical procedures) | 5 (5) | 0 (0)
Prostatectomy (Surgical and medical procedures) | 1 (1) | 2 (2)
Ptosis repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Radiotherapy (Surgical and medical procedures) | 2 (2) | 0 (0)
Radiotherapy to lung (Surgical and medical procedures) | 0 (0) | 1 (1)
Radiotherapy to rectum (Surgical and medical procedures) | 1 (1) | 0 (0)
Rectal prolapse repair (Surgical and medical procedures) | 2 (2) | 0 (0)
Removal of internal fixation (Surgical and medical procedures) | 1 (1) | 0 (0)
Renal stone removal (Surgical and medical procedures) | 1 (1) | 1 (1)
Resuscitation (Surgical and medical procedures) | 1 (1) | 5 (5)
Shoulder operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 4 (4) | 3 (3)
Small intestinal resection (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal decompression (Surgical and medical procedures) | 3 (3) | 0 (0)
Spinal laminectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal operation (Surgical and medical procedures) | 3 (3) | 4 (5)
Surgery (Surgical and medical procedures) | 2 (2) | 1 (1)
Therapeutic procedure (Surgical and medical procedures) | 16 (22) | 6 (7)
Thoracic cavity drainage (Surgical and medical procedures) | 2 (2) | 2 (3)
Thrombectomy (Surgical and medical procedures) | 2 (2) | 5 (5)
Thrombolysis (Surgical and medical procedures) | 0 (0) | 4 (4)
Thyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Toe amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Tracheostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Transcatheter aortic valve implantation (Surgical and medical procedures) | 6 (6) | 5 (5)
Transfusion (Surgical and medical procedures) | 58 (78) | 28 (37)
Transurethral bladder resection (Surgical and medical procedures) | 9 (11) | 4 (5)
Transurethral prostatectomy (Surgical and medical procedures) | 5 (5) | 2 (3)
Tumour excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Umbilical hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Ureteral stent insertion (Surgical and medical procedures) | 4 (4) | 2 (2)
Ureteral stent removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Urethrotomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Urinary cystectomy (Surgical and medical procedures) | 2 (2) | 0 (0)
Urinary incontinence surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Uterine prolapse repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Vaginal prolapse repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Varicose vein operation (Surgical and medical procedures) | 3 (3) | 0 (0)
Vascular operation (Surgical and medical procedures) | 2 (2) | 4 (5)
Vitrectomy (Surgical and medical procedures) | 1 (2) | 0 (0)
Vocal cord operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Angiodysplasia (Vascular disorders) | 5 (6) | 0 (0)
Aortic aneurysm (Vascular disorders) | 4 (5) | 0 (0)
Aortic stenosis (Vascular disorders) | 3 (3) | 2 (2)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Bleeding varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 4 (4)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1)
Giant cell arteritis (Vascular disorders) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 4 (4) | 3 (3)
Haemorrhage (Vascular disorders) | 18 (20) | 10 (10)
Hypertension (Vascular disorders) | 3 (3) | 4 (4)
Hypertensive crisis (Vascular disorders) | 3 (4) | 3 (3)
Hypertensive emergency (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 3 (6) | 4 (4)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 4 (4) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 7 (7) | 6 (8)
Peripheral artery occlusion (Vascular disorders) | 2 (3) | 2 (2)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 2 (2)
Peripheral embolism (Vascular disorders) | 1 (1) | 3 (3)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Thrombophlebitis (Vascular disorders) | 2 (2) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Venous stenosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edoxaban (N=1306) | ASA or Placebo (N=1302)
Anaemia (Blood and lymphatic system disorders) | 12 (13) | 8 (8)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
Lymph node calcification (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Angina pectoris (Cardiac disorders) | 12 (13) | 8 (10)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (6) | 11 (11)
Atrial flutter (Cardiac disorders) | 9 (10) | 4 (4)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 20 (29) | 18 (18)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial fibrosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 20 (20) | 7 (7)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 2 (3) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 6 (7) | 3 (3)
Auricular swelling (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 8 (9) | 7 (8)
Graves' disease (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 4 (4) | 3 (3)
Age-related macular degeneration (Eye disorders) | 1 (1) | 1 (1)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 9 (11) | 7 (8)
Cataract nuclear (Eye disorders) | 0 (0) | 1 (1)
Charles Bonnet syndrome (Eye disorders) | 0 (0) | 1 (1)
Choroidal haemorrhage (Eye disorders) | 2 (2) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 2 (2) | 2 (2)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Conjunctival irritation (Eye disorders) | 1 (1) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 1 (1) | 0 (0)
Dermatochalasis (Eye disorders) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 3 (3) | 3 (3)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 3 (3) | 0 (0)
Eyelid bleeding (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 2 (3)
Macular degeneration (Eye disorders) | 1 (1) | 1 (1)
Maculopathy (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 2 (2) | 1 (1)
Optic disc haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 1 (1)
Visual acuity reduced (Eye disorders) | 2 (2) | 0 (0)
Visual impairment (Eye disorders) | 3 (8) | 5 (5)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 16 (19)
Abdominal pain upper (Gastrointestinal disorders) | 10 (10) | 3 (3)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (5) | 8 (8)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 19 (20) | 20 (21)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 3 (3)
Flatulence (Gastrointestinal disorders) | 1 (1) | 2 (2)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 7 (7) | 8 (8)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 7 (7) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 3 (5) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lip haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 2 (2) | 2 (2)
Mouth haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 21 (21) | 11 (11)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Peritoneal cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 9 (9) | 5 (6)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2) | 2 (2)
Trichoglossia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 5 (5)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 18 (20) | 15 (17)
Chest discomfort (General disorders) | 2 (2) | 1 (1)
Chest pain (General disorders) | 20 (21) | 19 (20)
Complication associated with device (General disorders) | 2 (2) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 8 (8) | 11 (11)
Gait disturbance (General disorders) | 2 (2) | 4 (4)
General physical health deterioration (General disorders) | 3 (3) | 2 (2)
Illness (General disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 10 (10) | 4 (4)
Non-cardiac chest pain (General disorders) | 7 (13) | 7 (7)
Oedema (General disorders) | 6 (6) | 3 (3)
Oedema peripheral (General disorders) | 16 (20) | 19 (19)
Pain (General disorders) | 3 (3) | 0 (0)
Peripheral swelling (General disorders) | 7 (7) | 7 (7)
Pyrexia (General disorders) | 4 (4) | 5 (5)
Swelling face (General disorders) | 1 (1) | 0 (0)
Ulcer (General disorders) | 1 (1) | 0 (0)
Vaccination site haematoma (General disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Congestive hepatopathy (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Primary biliary cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 5 (5) | 7 (7)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (3) | 1 (2)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 6 (6) | 2 (2)
Cystitis (Infections and infestations) | 5 (6) | 2 (2)
Dacryocystitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 1 (1)
Ear infection (Infections and infestations) | 3 (4) | 0 (0)
Ear infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 2 (2) | 2 (2)
Eye infection (Infections and infestations) | 0 (0) | 1 (2)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 2 (2)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 3 (3)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 2 (2) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 6 (8)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 6 (6) | 11 (11)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 4 (4)
Pulpitis dental (Infections and infestations) | 1 (4) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 6 (6) | 8 (11)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 2 (2) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 5 (5)
Urinary tract infection (Infections and infestations) | 18 (33) | 19 (24)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 2 (3)
Accidental overdose (Injury, poisoning and procedural complications) | 4 (5) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Bone fissure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 8 (8) | 4 (4)
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eyelid injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 32 (37) | 31 (35)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 4 (5) | 13 (13)
Heat exhaustion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 6 (6)
Implantation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 5 (7) | 7 (8)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shoulder fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Silicosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Skin laceration (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Angiocardiogram (Investigations) | 2 (2) | 1 (1)
Angiogram (Investigations) | 2 (2) | 0 (0)
Arthroscopy (Investigations) | 0 (0) | 1 (1)
Biopsy intestine (Investigations) | 1 (1) | 0 (0)
Biopsy lymph gland (Investigations) | 0 (0) | 2 (2)
Biopsy prostate (Investigations) | 2 (2) | 1 (1)
Bleeding time prolonged (Investigations) | 4 (4) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 1 (1)
Bronchial aspiration procedure (Investigations) | 1 (1) | 0 (0)
Bronchoscopy abnormal (Investigations) | 0 (0) | 1 (1)
Catheterisation cardiac (Investigations) | 3 (3) | 1 (1)
Colonoscopy (Investigations) | 5 (5) | 2 (2)
Coronavirus test positive (Investigations) | 48 (49) | 30 (30)
Cystoscopy (Investigations) | 0 (0) | 1 (1)
Dental examination (Investigations) | 0 (0) | 1 (1)
Diagnostic procedure (Investigations) | 1 (1) | 0 (0)
Echocardiogram (Investigations) | 0 (0) | 1 (1)
Echocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 2 (2)
Endoscopy (Investigations) | 1 (1) | 0 (0)
Endoscopy upper gastrointestinal tract (Investigations) | 2 (2) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0)
Glomerular filtration rate increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin increased (Investigations) | 0 (0) | 1 (1)
Heart rate decreased (Investigations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 3 (3)
International normalised ratio abnormal (Investigations) | 0 (0) | 1 (1)
Low density lipoprotein increased (Investigations) | 0 (0) | 1 (1)
Magnetic resonance imaging (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1 (1) | 1 (1)
Radioisotope scan (Investigations) | 0 (0) | 1 (1)
Rectal ultrasound (Investigations) | 0 (0) | 1 (1)
Serum ferritin decreased (Investigations) | 0 (0) | 1 (1)
Sleep study (Investigations) | 1 (1) | 0 (0)
Spirometry (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Vitamin D decreased (Investigations) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 5 (5) | 7 (8)
Weight increased (Investigations) | 2 (2) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 7 (7) | 4 (4)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (23) | 24 (27)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 19 (25)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint microhaemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (10) | 3 (4)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (9) | 15 (16)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Vertebral lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (3)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Colorectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 5 (5)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (3)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Axonal neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 2 (2)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 3 (3) | 5 (5)
Dementia (Nervous system disorders) | 3 (3) | 6 (6)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 47 (57) | 46 (52)
Dizziness postural (Nervous system disorders) | 1 (1) | 2 (2)
Dysarthria (Nervous system disorders) | 0 (0) | 2 (2)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 20 (21) | 19 (21)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 2 (2)
Memory impairment (Nervous system disorders) | 1 (2) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Ophthalmic migraine (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 6 (6) | 2 (2)
Parkinson's disease (Nervous system disorders) | 1 (1) | 3 (3)
Polyneuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 3 (3) | 5 (5)
Seizure (Nervous system disorders) | 1 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 15 (16) | 11 (14)
Tremor (Nervous system disorders) | 1 (1) | 2 (2)
Vascular dementia (Nervous system disorders) | 0 (0) | 2 (3)
Device electrical impedance issue (Product Issues) | 0 (0) | 1 (1)
Device inappropriate shock delivery (Product Issues) | 0 (0) | 1 (1)
Device lead damage (Product Issues) | 0 (0) | 1 (1)
Device lead issue (Product Issues) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Device stimulation issue (Product Issues) | 1 (2) | 0 (0)
Lead dislodgement (Product Issues) | 0 (0) | 1 (1)
Thrombosis in device (Product Issues) | 0 (0) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (4) | 4 (4)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Apathy (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 3 (3)
Depressed mood (Psychiatric disorders) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 4 (4) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 1 (1)
Bladder wall calcification (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 5 (6) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (4) | 1 (1)
Haematuria (Renal and urinary disorders) | 31 (41) | 8 (10)
Nocturia (Renal and urinary disorders) | 1 (1) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 8 (8)
Diaphragmatic spasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 43 (46) | 42 (50)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 48 (54) | 21 (22)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Chronic papillomatous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (13) | 8 (8)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 10 (11) | 9 (12)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Breast prosthesis user (Social circumstances) | 1 (1) | 0 (0)
Living in residential institution (Social circumstances) | 0 (0) | 1 (1)
Arthrodesis (Surgical and medical procedures) | 1 (1) | 0 (0)
Bladder neoplasm surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Blepharoplasty (Surgical and medical procedures) | 0 (0) | 2 (2)
Bunion operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Cancer surgery (Surgical and medical procedures) | 1 (1) | 3 (3)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac pacemaker removal (Surgical and medical procedures) | 1 (1) | 1 (1)
Cardiac pacemaker replacement (Surgical and medical procedures) | 36 (36) | 39 (40)
Cardiac resynchronisation therapy (Surgical and medical procedures) | 6 (6) | 3 (3)
Cardioversion (Surgical and medical procedures) | 6 (7) | 9 (11)
Carpal tunnel decompression (Surgical and medical procedures) | 3 (3) | 3 (3)
Cataract operation (Surgical and medical procedures) | 11 (15) | 12 (15)
Catheter management (Surgical and medical procedures) | 0 (0) | 2 (3)
Cholelithotomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Dental implantation (Surgical and medical procedures) | 1 (1) | 0 (0)
Electrocauterisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Eye operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Eyelid operation (Surgical and medical procedures) | 2 (4) | 0 (0)
Finger amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastric polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Haematoma evacuation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Hydrocele operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Internal fixation of fracture (Surgical and medical procedures) | 0 (0) | 1 (1)
Jaw operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee operation (Surgical and medical procedures) | 1 (1) | 2 (3)
Large intestinal polypectomy (Surgical and medical procedures) | 5 (5) | 0 (0)
Liver operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Medical device removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Mole excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Papilloma excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Percutaneous coronary intervention (Surgical and medical procedures) | 1 (1) | 1 (1)
Peripheral artery angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Prostatic operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Radiotherapy to prostate (Surgical and medical procedures) | 1 (1) | 1 (1)
Rhinoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Rhizolysis (Surgical and medical procedures) | 1 (1) | 0 (0)
Sclerotherapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Shoulder operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin lesion removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 8 (10) | 5 (6)
Skin operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Toe amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 11 (12) | 4 (4)
Transurethral bladder resection (Surgical and medical procedures) | 0 (0) | 1 (1)
Angiodysplasia (Vascular disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 3 (3) | 2 (2)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Aortic dilatation (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Aortic thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Bleeding varicose vein (Vascular disorders) | 2 (2) | 0 (0)
Blood pressure fluctuation (Vascular disorders) | 1 (1) | 2 (2)
Circulatory collapse (Vascular disorders) | 2 (2) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 21 (24) | 17 (17)
Haemorrhage (Vascular disorders) | 4 (6) | 2 (2)
Hot flush (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 8 (8) | 10 (11)
Hypertensive crisis (Vascular disorders) | 4 (4) | 4 (4)
Hypertensive emergency (Vascular disorders) | 0 (0) | 3 (3)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 13 (14) | 11 (12)
Intermittent claudication (Vascular disorders) | 2 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 4 (4) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 2 (2)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral venous disease (Vascular disorders) | 2 (3) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 1 (1)
Subgaleal haematoma (Vascular disorders) | 0 (0) | 1 (1)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Thrombophlebitis (Vascular disorders) | 1 (1) | 2 (2)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Varicose ulceration (Vascular disorders) | 1 (1) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial does not have sufficient power to detect or rule out a small beneficial effect of oral anticoagulation on the prevention of stroke. The generalizability of these findings with edoxaban to other NOACs is not known.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT02618577/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT02618577/SAP_001.pdf